CLINICAL TRIAL: NCT05894915
Title: Study and Transformation of Tumor Molecular Features Screening Model of Endometrial Carcinoma Surgical Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Wang, Chief Physician, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022PHB105-002
Record Dates: First submitted 2023-04-29; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Endometrial Carcinoma; Tumor Molecular Features Screening Model
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open surgery group (Experimental): Patients who met the inclusion criteria and excluded the exclusion criteria, and did not have high mutational burden characteristics after molecular testing, were randomly divided into open surgery group or laparoscopic surgery group according to 1:1.
  Interventions: Procedure: open surgery
- laparoscopic surgery group (Experimental): Patients who met the inclusion criteria and excluded the exclusion criteria, and did not have high mutational burden characteristics after molecular testing, were randomly divided into open surgery group or laparoscopic surgery group according to 1:1.
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: open surgery — Open surgery is a traditional surgery method.
  Arms: open surgery group
Procedure: laparoscopic surgery — Laparoscopic surgery is a newly developed minimally invasive method.
  Arms: laparoscopic surgery group

SUMMARY:
At present, endometrial carcinoma is one of the three most common malignant tumors in gynecology, and the incidence has been increasing year by year, causing a large health and economic burden to the society. Therefore, researchers regard the hierarchical management and precise diagnosis and treatment of endometrial carcinoma as an important direction for future research. In 2013, the American Cancer Genome Atlas Research Network proposed a molecular typing of endometrial carcinoma. In recent years, international scholars have conducted relevant research on the molecular characteristics of a large number of endometrial carcinomas and immunity, targeted therapy and postoperative adjuvant chemoradiotherapy. However, the molecular characteristics of endometrial carcinoma and the choice of surgical route are still in a relatively lacking state. The previous research of the investigators' group was the first to propose the concept of selecting surgical routes for endometrial carcinoma based on molecular characteristics. Then, on this basis, the investigators' research group plans to carry out a prospective randomized controlled study to further analyze the impact of surgical routes on the short-term safety and long-term prognosis of endometrial carcinoma patients with different molecular characteristics, and transform it into a clinical decision-making technical index system for endometrial carcinoma surgical selection based on molecular characteristics and further promote and apply. The results of this study will make up for the shortcomings in the relevant fields of endometrial carcinoma research in the world to some extent, and become an important aspect of the decision-making system of clinical comprehensive precision diagnosis and treatment of endometrial carcinoma patients.

DETAILED DESCRIPTION:
1. Research purpose and significance Endometrial carcinoma is one of the three most common malignant tumors in gynecological diseases. At present, its emergence has caused a relatively serious health economic burden worldwide, according to statistics, the number of new cases of endometrial carcinoma in the world exceeded 400,000 in 2020. In China, the incidence of endometrial carcinoma is second only to cervical cancer and ranks second among female reproductive tract malignancies. In recent years, public health problems such hypertension, diabetes mellitus and poor lifestyle have become increasingly serious, which has led to an increase in the incidence of endometrial carcinoma and a younger age of onset.

   The prognosis of patients with endometrial carcinoma is closely related to their clinicopathological features, such as stage, grade, and pathological subtype. Stratified individualized diagnosis and treatment of endometrial carcinoma patients is an important direction that international scholars have been constantly exploring. In 1983, Bohkman proposed the dichotomous classification systemof endometrial carcinoma, which is based on the pathological characteristics to divide endometrial carcinoma into two types, type I carcinoma into two types, of which type I cancer mainly refers to endometrioid adenocarcinoma, type II carcinoma includes serous carcinoma, clear cell carcinoma and other special types. However, further evidence suggests that this approach is still limited in guiding patients' management and outcome. In 2013, American scholars used he Cancer Genome Atlas data to further propose the molecular typing of endometrial carcinoma, which divided endometrial carcinoma into four categories: POLE (ultramutated)，microsatellite instability (MSI)hypermutated, Copy-number low(CNL) and Copy-number high(CNH). Among them, POLE (ultramutated)type has the best prognosis, CNH type has the worst prognosis, and the other two types are in the middle. Effective individualized diagnosis and treatment according to the clinicopathological and molecular characteristics of patients is a hot issue that international scholars are concerned about and is of great significance. At present, there are clinical trials related to postoperative adjuvant therapy based on molecular characteristics, and a large number of studies on targeted therapy and immunotherapy support the clinical application of related drugs，so far, research on molecular characteristics and endometrial carcinoma surgery is still in a state of scarcity.

   In 2018, American scholars published a prospective and retrospective study on laparoscopic surgery for the treatment of early cervical carcinoma. The results suggest that the risk of recurrence and death in the minimally invasive surgery group is much higher than in the open surgery group, and the reasons are likely to include uterine lifting cup, the effects of laparoscopic CO2 pneumoperitoneum, or surgeon experience. It led the investigators to wonder whether similar factors would also have an impact on the safety of eminimally invasive surgery in endometrial carcinoma. Furthermore, regarding the choice of the endometrial carcinoma surgical route, although large-scale clinical trials have demonstrated that the prognosis of patients after minimally invasive surgery and open surgery is similar, the current study did not include patient molecular characteristics. According to the clinicopathological and molecular characteristics of patients, the formulation of personalized surgical strategies suitable for different groups of people is an important clinical problem that needs to be solved urgently.

   This project is based on theresults of previous retrospective studies of this research group, so as to carry out prospective randomized controlled studies, further evaluate the impact of surgical approaches on the prognosis of patients with endometrial cancer with different molecular characteristics, establish a clinical application model based on molecular characteristics to guide the selection of surgical routes, and transform it into a clinical decision-making technical index system for endometrial cancer surgical selection based on molecular characteristics for further promotion and application.
2. The research status at home and abroad After TCGA endometrial carcinoma molecular typing was proposed in 2013, many international research teams further simplified it, which greatly promoted the clinical promotion and application of molecular typing. The existing endometrial carcinoma typing system includes the PromisE classification proposed by Canadian scholars, TranPORTEC typing proposed by Dutch scholars. Based on this, the researchers carried out further work on molecular characteristics to guide patients with postoperative adjuvant therapy. Recently, Dutch scholars have further analyzed the effects of different molecular characteristics on the efficacy of adjuvant chemoradiotherapy in high-risk endometrial carcinoma patients based on PORTEC3 research data ，and are designing a prospective randomized controlled trial (i.e., PORTEC-4a study) based on TransPORTEC classification guidance for postoperative adjuvant radiotherapy in patients with high-risk endometrial carcinoma. Recently, Korean scholars published an analysis on the efficacy of PromisE typing and fertility preserving treatment of endometrial cancer. The above studies show that patients with different molecular characteristics respond differently to different therapeutic measures, so further establishing individualized diagnosis and treatment strategies for patients with different subtypes is an important direction for future research.

   Surgery is the most important part of the endometrial carcinoma complex. Moreover, the application of minimally invasive techniques significantly reduced the incidence of perioperative complications, reduced intraoperative blood loss, and shortened the average length of hospital stay，but the long-term safety of this technique is still an important issue worthy of further investigation. Although clinical trials have confirmed that the long-term prognosis of minimally invasive surgery for early endometrial carcinoma is similar to that of open surgery，none of the above studies included the molecular characteristics of patients. In recent years, more and more research evidence has shown the importance of molecular characteristics in the prognosis and stratified management of endometrial carcinoma patients, so it is necessary to further evaluate and analyze the prognosis of endometrial carcinoma patients with different molecular characteristics after minimally invasive surgery.

   Since 2018, American scholars proposed that laparoscopic radical hysterectomy is associated with poor prognosis in patients with early cervical cancer compared with open surgery, research teams in various countries have carried out further research and analysis on the relationship between surgical methods and the long-term prognosis of cervical cancer patients, and most of the conclusions are consistent with the results of American scholars. A recent meta-analysis pooled the results of 15 clinical studies and further confirmed the adverse effects of minimally invasive surgery on the prognosis of cervical cancer patients. The above research has led us to further think about this question, that is, the endometrial carcinoma laparoscopic surgery also has the influence of pneumoperitoneum, uterine cup and other factors, so is it also associated with a poorer prognosis?This issue needs to be further examined and analyzed. Recently, on the basis of large-scale retrospective analysis, scholars have put forward the view that the use of uterine cups in laparoscopic surgery is related to the adverse prognosis of patients with endometrial carcinoma, and the possible mechanism of uterine cups promoting intraperitoneal spread has been further elaborated. Furthermore, a recent study by Canadian scholars suggested that the disease-free survival of patients with endometrial carcinoma after robotic-assisted laparoscopic surgery was significantly shortened, and suggested that this situation is most likely related to the delay in postoperative adjuvant radiotherapy caused by delayed healing of the vaginal cuff after minimally invasive surgery. According to the above situation, more and more evidences suggests that the investigators still need to conduct a more in-depth and detailed analysis of the safety of laparoscopic surgery in the treatment of endometrial carcinoma, and further analyze the prognostic impact of different surgical methods based on molecular characteristics, which is of great significance to the establishment of a precise individualized diagnosis and treatment system of endometrial carcinoma in the future.
3. The preliminary research results directly related to this project support the research team Based on the retrospective TCGA data, the research team analyzed the effect of surgical pathway on the prognosis of endometrial carcinoma patients with different molecular characteristics. According to preliminary studies, patients with MSI endometrial carcinoma who underwent minimally invasive and had similar prognosis after laparotomy, while patients with microsatellite stability endometrial carcinoma who underwent minimally invasive surgery had significantly shorter recurrence-free survival than those in the open surgery group. Therefore, the investigators believe that MSI endometrial carcinoma has a higher mutational load and can promote neoantigen expression, resulting in a stronger anti-tumor immune response in vivo, which may balance the negative effects of laparoscopic surgery in promoting tumor dissemination, but this feature is not present in microsatellite stability tumors.

Subsequently, the investigators further analyzed the relationship between other molecular features and the prognosis of patients with endometrial carcinoma undergoing different surgical procedures. According to the investigators' study, endometrial carcinoma patients with POLE gene mutations, homologous recombinant repair pathway mutations, and MUC16 gene mutations had a similar prognosis after minimally invasive surgery than the open surgery group, while patients with TP53 gene mutations had significantly shorter recurrence-free survival after minimally invasive surgery than those in the open surgery group. Through the above results, the investigators preliminarily established an Endometrial Carcinoma selection model based on molecular features. The above research results have laid a solid foundation for the investigators' further prospective clinical research and serve as strong support for this study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-80 years.
* Preoperative hysteroscopic biopsy pathology is endometrial carcinoma, preoperative imaging evaluation of tumor limited to uterine or extrauterine metastasis limited to pelvic or para-aortic lymph nodes.
* No liver and kidney function abnormalities and bone marrow suppression before surgery.
* ECOG score 0 points.
* Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.
* Molecular testing has confirmed that the participant does not have high mutational burden characteristics (including POLE mutations, MSI-H, homologous recombinant repair pathway mutations).

Exclusion Criteria:

* Preoperative adjuvant therapy.
* Have contraindications to chemoradiotherapy and cannot receive postoperative adjuvant chemoradiotherapy.
* Previous history of other malignant tumors or other malignant tumors at the same time.
* Laparoscopic surgery transferred to open surgery for special reasons.
* unable or unwilling to comply with the requirements of the study.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 390 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence rate of each group | 2 year
  the proportion of radiographic or pathologically confirmed recurrence cases to the total number of cases in this group up to 2-year follow-up.

SECONDARY OUTCOMES:
time of the surgery process | 1 day
intraoperative blood loss | 1 day
  use hematocrit method or gauze weighing method to estimate the intraoperative blood loss.
Complication rate within 8 weeks after surgery | 8weeks
  Follow-up plan: patients are followed up regularly after surgery for suspicious signs of Complication.
average length of hospital stay | 1 month
Tumor recurrence time | 2 year
  Follow-up plan: patients are followed up regularly after surgery for signs of recurrence.
Tumor recurrence site | 2year
  Follow-up plan: patients are followed up regularly after surgery for suspicious signs of recurrence.
no recurrence survival | 5 year
  Follow-up plan: patients are followed up regularly after surgery for suspicious signs of recurrence.
Overall lifetime survival | 5 year
  Follow-up plan: patients are followed up regularly after surgery (every 3 months from the end of chemoradiotherapy). Follow-up includes the patient's symptoms, By phone call or WeChat mini program to find if there are suspicious signs of recurrence.

IPD SHARING:
Plan to Share IPD: No